CLINICAL TRIAL: NCT01122550
Title: Reproducibility Study of OABSS and Its Response to Treatment in Indonesia - Part 1: Reproducibility -
Brief Title: Reproducibility Study of Overactive Bladder Symptom Score [OABSS]
Acronym: RESORT-1
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Indonesia Inc. (Industry)
Responsible Party: Disclosure Director, Astellas Pharma, Inc
Other Study IDs: EQL-CRU.004-2009
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Overactive Bladder
Keywords: OABSS; IPSS; PPBC; 3-day micturition diary
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate its reproducibility of overactive bladder symptom score (OABSS) and to evaluate its correlation to other measures of OAB symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms OAB for 3 months or longer
* At least 1 urgency episode in last 3 days
* Symptoms of OAB as verified by 3-day micturition diary prior to Visit 1, defined by:

  * Number of micturition per day ≥8
  * Number of urgency episodes in 3 days ≥1

Exclusion Criteria:

* Significant stress incontinence or mixed stress/urge incontinence
* Subjects with indwelling catheters or practicing intermittent self-catheterization
* Symptomatic urinary tract infection, chronic inflammation
* Diabetic neuropathy
* Drug or non-drug treatment for OAB was started, quitted or changed in 4 weeks
* Participation in any clinical trial in 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic OAB patients having urgency episodes
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
OABSS | Weeks 0 and 2

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) | Weeks 0 and 2
Quality of Life (QOL) score | Weeks 0 and 2
Patient Perception of Bladder Condition (PPBC) | Weeks 0 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Indonesia
Locations (3):
- Indonesia (3):
  - Bandung
  - Jakarta
  - Surabaya